CLINICAL TRIAL: NCT04097171
Title: The Effect of Diet Composition on Performance, Energy Expenditure, Blood Lipids and Lipoproteins, and Cognitive Function and Mood States in Highly Trained Cyclists
Brief Title: The Effect of Diet Composition on Performance, Expenditure, Blood Lipids, and Appetite Hormones in Highly Trained Cyclists
Acronym: DCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Meena Shah, Interim Chair, Professor and Director, Graduate Program, Texas Christian University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CT2019MS3
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Endurance Cycling Performance
MeSH Terms: interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Carbohydrate Diet (Experimental): Participants will consume a high carbohydrate diet (65-75% of total energy intake). Protein intake will be standardized at 15% of total energy intake.
  Interventions: Other: Diet
- Ketogenic Diet (Experimental): Participants will consume a low carbohydrate diet (<5-10% of total energy intake). Protein intake will be standardized at 15% of total energy intake.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Participants will consume each diet for 14 days in a crossover design.

SUMMARY:
This study employs a crossover design to evaluate the effect of two different diets (high carbohydrate vs. ketogenic) and corresponding test meals on endurance exercise performance, energy expenditure including resting metabolic rate and thermic effect of food, postprandial responses of blood lipids, glucose and appetite hormones, and cognitive function and mood states.

DETAILED DESCRIPTION:
Traditionally, a high carbohydrate diet is recommended for elite endurance athletes and sub-elite, highly trained recreational athletes competing in endurance events. However, recently the ketogenic diet (extremely low carbohydrate content) has become popular in these populations. The effect on endurance exercise performance, energy expenditure, postprandial blood profiles, and cognitive function and mood states requires further investigation.

In this study, highly trained recreational cyclists and triathletes will adhere to each diet (high-carbohydrate and ketogenic) for 14 days in a crossover design. Experimental trials at baseline and after each diet will evaluate endurance cycling performance (time trial), resting energy expenditure, the thermic effect of food of test meals corresponding in composition to each diet, postprandial responses of blood lipids, glucose and appetite hormones, and cognitive function and mood states.

ELIGIBILITY:
Inclusion Criteria:

* >100-150km of cycling per week
* VO2max > 80th percentile for sex and age (adjusted for cycle ergometry)
* apparently healthy

Exclusion Criteria:

* weight loss supplements/medications/diet
* extreme dietary patterns (e.g. extremely high or low carbohydrate)
* nicotine use
* heavy alcohol use (>7 drinks/week female; >14 drinks/week male)
* food allergies
* diabetes
* heart disease
* stroke
* liver/kidney/thyroid disease
* anemia
* eating disorders
* uncontrolled hypertension
* pulmonary/orthopedic/musculoskeletal problems that prevent exercise
* surgery that affects swallowing and digestion
* claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Endurance Cycling Performance | 180 min after the meal begins
  Time to completion in a 30-kilometer simulated time trial

SECONDARY OUTCOMES:
Respiratory Exchange Ratio | Change from baseline at 30 min, 60 min, 90 min, 120 min, 150 min, 180 min, 192 min, 204 min, 216 min, 228 min and 240 min after the meal begins
  Indirect calorimetry fasted, postprandial, and during exercise
Muscle Fuel Rating | Change from baseline at 180 min and 240 min after the meal begins
  Ultrasound echogenicity of Rectus Femoris
Oxygen consumption (VO2) | At 192 min, 204 min, 216 min, 228 min and 240 min after the meal begins
  Indirect calorimetry during exercise
Rating of Perceived Exertion (RPE) | At 192 min, 204 min, 216 min, 228 min and 240 min after the meal begins
  6-20 Borg's scale during exercise
Thermic Effect of Food (postprandial energy expenditure) | Change from baseline at 30 min, 60 min, 90 min, 120 min, 150 min, 180 min after the meal begins
  Fasted vs. postprandial indirect calorimetry
Subjective appetite ratings | Change from baseline at 60 min, 120 min, 180 min after the meal begins
  Visual Analog Scale (Scale 1: Perception of Hunger [0-100 mm]; Scale 2: Perception of Fullness [0-100 mm]; Scale 3: Desire to Eat [0-100 mm]
Appetite hormones including ghrelin, leptin, insulin, and Peptide-YY | Change from baseline at 30 min, 60 min, 120 min, 180 min and 240 min
  Fasted, postprandial & post exercise blood concentration of appetite hormones
Blood glucose | Change from baseline at 180 min and 240 min after the meal begins; on day 7 of each diet
  Fasted, postprandial & post exercise blood concentration of glucose
Blood pressure | Change from baseline at 180 min after the meal begins
  Fasted, postprandial & post exercise
Cognitive function | At 180 min and 240 min after the meal begins
  Stroop test
Mood state questionnaire | At 180 min and 240 min after the meal begins
  Abbreviated Profile of Mood States; 40-item scale; Likert scale from 0 = "not at all" to 4 = "extremely"
Resting Metabolic Rate | At baseline before meal begins
  Indirect calorimetry in fasted state
Blood lipids including (triglycerides, total cholesterol, low density lipoprotein, and high-density lipoprotein) | Change from baseline at 30 min, 60 min, 120 min, 180 min, 192 min, 204 min, 216 min, 228 min and 240 min after the meal begins
  Fasted and postprandial in mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data of all outcome variables will be shared on an Open Science Framework project page (osf.io) along with the study protocol, statistical analysis plan, and analytic code
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Will become available at the latest June 2021 and be available indefinitely
Access Criteria: Openly available
URL: http://osf.io/ujx6e/

REFERENCES:
- [Derived] Graybeal AJ, Kreutzer A, Moss K, Shah M. Changes in the chronic and postprandial blood lipid profiles of trained competitive cyclists and triathletes following a ketogenic diet: a randomized crossover trial. BMC Sports Sci Med Rehabil. 2024 Jan 16;16(1):19. doi: 10.1186/s13102-023-00801-5. PMID 38229197